CLINICAL TRIAL: NCT02875327
Title: Linkage of Medicaid Enrollment Lnformation to Surveillance, Epidemiology and End Results Data
Brief Title: Linkage of Medicaid Enrollment Information to Surveillance, Epidemiology and End Results Data
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916163; 16-C-N163
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Neoplasm; Health Services Accessibility; Outcome Assessment; Healthcare Disparities
Keywords: SEER; Medicaid; Cancer; Health Services Research; Epidemiology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

SUMMARY:
Background:

The SEER database collects data about people with cancer. SEER stands for Surveillance, Epidemiology, and End Results. Medicaid is a kind of health insurance. It is for people who have low income or serious medical needs. Many studies have shown that Medicaid recipients with cancer are more likely to be diagnosed later in the disease than people with other insurance. They are also less likely to get treatment. Researchers want to compare Medicaid data and SEER data. They want to make this available to other scientists.

Objectives:

To link people in the SEER database to Medicaid data for the years around their cancer diagnosis. To create a file that contains SEER case numbers linked to Medicaid numbers.

Eligibility:

No people are enrolled in this study.

Design:

The SEER finder file will be securely uploaded to the CMS Data Center.

The finder file will be matched against the Medicaid Personal Summary file at the CMS Data Center.

If participants appear in both the SEER file and Medicaid file, their data will be extracted.

The dates of Medicaid data will be compared with the SEER date of diagnosis. Researchers will see if the Medicaid dates fall in certain periods. These are 12 months before, the month of, and 11 months after diagnosis.

If participants are eligible for Medicaid for these periods, a flag will be created in the file. It will note the participants is eligible and why.

The SEER finder file will be destroyed.

The only data saved will be:

Each participant's unique random SEER case number linked to their Medicaid number

Monthly flags about Medicaid eligibility

DETAILED DESCRIPTION:
Numerous studies have demonstrated that Medicaid recipients with cancer are more likely to be diagnosed at an advance stage and less likely to receive recommended treatment than are patients with other types of health insurance. The objective of this project is to link persons included in the Surveillance, Epidemiology and End Results (SEER) data to Medicaid enrollment information during the year before and after their cancer diagnosis. NCI is also seeking permission to create and maintain a file that crosswalks each patient's SEER case number to their Medicaid enrollment number. Information about Medicaid enrollment would be available by special request to all researchers who want to use SEER data to assess the impact of Medicaid enrollment on stage and treatment.

ELIGIBILITY:
* INCLUSION:
* Cancer Diagnosis
* Medicaid Member
* Registered within the SEER Program

EXCLUSION:

-None

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medicaid beneficiaries diagnosed with cancer living in the SEER cancer registry catchment areas.
Sampling Method: Non-Probability Sample
Enrollment: 3217145 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Link persons included in the Surveillance, Epidemiology and End Results (SEER) data to Medicaid enrollment information | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey R Enewold, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Derived] Huang J, Shi H, Ge L, Zhu B, Liu J, Wang X, Han Z, Li Q, Wang Z. Epidemiologic and survival analysis of malignant peripheral nerve sheath tumors: a retrospective cohort study. Int J Surg. 2024 Dec 1;110(12):8210-8214. doi: 10.1097/JS9.0000000000001756. No abstract available. PMID 38935102